CLINICAL TRIAL: NCT04801368
Title: A Randomized-Controlled Trial Comparing Long-acting and Short-acting Local Anesthetics at the Time of Penile Prosthesis Placement
Brief Title: Randomized Trial of Ropivacaine & Bupivacaine for Inflatable Penile Prosthesis
Acronym: ROVEX-IPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew (Matt) J. Ziegelmann, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20-010842
Record Dates: First submitted 2021-02-19; First posted 2021-03-17 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: The two anesthetics being used in the study are FDA approved and used in standard practice for the procedure. Subjects will be blindly assigned to one of two study groups at the initial phase of the study.
Who Masked: Participant
Masking Description: Patient is blind to local anesthetic being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Receiving Ropivacaine (Experimental): Patients receiving Ropivacaine.
  Interventions: Drug: Randomization of two local anesthetics.
- Receiving Liposomal Bupivacaine (Experimental): Patients receiving Liposomal Bupivacaine.
  Interventions: Drug: Randomization of two local anesthetics.

INTERVENTIONS:
Drug: Randomization of two local anesthetics. — Patients will be blinded and randomized to two different arms. One receiving ropivacaine, one receiving liposomal bupivacaine.

SUMMARY:
The purpose of this research is to determine the effects of penile ring block for local anesthesia with liposomal bupivacaine vs ropivacaine mixture in subjects undergoing surgery for Penile Prosthesis Placement.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing 3-piece penile prosthesis placement under general anesthesia at Mayo Clinic - Rochester.
* ≥ 18 years old.

Exclusion Criteria:

* History of opioid exposure within the preceding 90 days prior to surgery (based on patient-report, review of the electronic medical record, and NMP prescribing database review)
* Current or prior history of alcohol or drug abuse (illicit or prescription)
* History of chronic pain conditions (chronic musculoskeletal pain, fibromyalgia, central sensitization, chronic pelvic pain syndrome, etc.)
* History of cardiac arrhythmia or untreated severe cardiovascular disease
* Uncontrolled hypertension
* Hepatic insufficiency
* Renal insufficiency (CKD stage IIIa or greater)
* Current anti-platelet or anti-coagulation therapy with plans to continue at the time of prosthesis placement
* Poorly controlled diabetes mellitus (defined as HgbA1c > 8.5 within 30 days of surgery)
* Concurrent adjunctive operative procedures planned at the time of penile prosthesis placement (examples: male urethral sling, Peyronie's disease straightening with penile plication or incision/grafting)
* Concurrent non-prosthetic surgery planned at the time of penile prosthesis placement (examples: circumcision, hernia repair, hydrocelectomy, etc.)
* Planned infrapubic or subcoronal incision at the time of penile prosthesis placement
* Patients who will be undergoing prosthesis placement using local, monitored, or spinal anesthesia (i.e. non-general anesthesia)
* Allergy or history of intolerance to any local anesthetic agents included in the protocol
* History of prior penile prosthesis or artificial urinary sphincter surgery
* Revision penile prosthesis surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Ziegelmann, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Receiving Ropivacaine: Patients receiving Ropivacaine intra-operatively.
  Randomization of two local anesthetics.: Patients will be blinded and randomized to two different arms. One receiving ropivacaine, one receiving liposomal bupivacaine.
  Dosage depends on subjects height, weight, and other health factors
- Receiving Liposomal Bupivacaine: Patients receiving Liposomal Bupivacaine intra-operatively.
  Randomization of two local anesthetics.: Patients will be blinded and randomized to two different arms. One receiving ropivacaine, one receiving liposomal bupivacaine.
  Dosage depends on subjects height, weight, and other health factors
Period: Overall Study
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Started | 6 | 14
Completed | 5 | 14
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine | Total
Number analyzed (Participants) | 5 | 14 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10
  >=65 years | 2 | 7 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 14 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 13 | 17
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 12 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 14 | 19
State Trait Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — The State-Trait Anxiety Inventory (STAI) is a survey that measures a person's tendency to experience anxiety when faced with stress. Results are reported as units on a scale, minimum 20 (scoring low on a tendency to experience anxiety when faced with stress) to maximum of 80 (scoring high on a tendency to experience anxiety when faced with stress).
  Results may impact a subject's tendency to score higher on later measures, hence why this scale is used at a baseline visit.
  units on a scale | 27 (12.96) | 30.3 (11.24) | 29.39 (11.44)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: units on a scale] — The Pain Catastrophizing Scale is a questionnaire that measures how much someone catastrophizes about pain. Results are reported as units on a scale, minimum 0 (scoring low on a tendency to catastrophize pain, or rate pain as more tolerable than other people) to maximum of 52 (scoring high on a tendency to catastrophize pain, or rate pain as less tolerable than other people).
  Results may impact a subject's tendency to score higher on later pain measures, hence why this scale is used at a baseline visit.
  units on a scale | 1.6 (2.07) | 4.08 (5.75) | 3.39 (5.07)

OUTCOME MEASURES:

1. Primary Outcome: Visual-analogue Pain Scale
Description: Visual-analogue pain scale is a tool used to measure pain intensity at a specific timepoint, asking a patient to use visuals to rate their pain on a scale of 1 to 10.
  Results are reported as units on a scale, minimum 1 (experiencing the least amount of pain possible) to maximum of 10 (experiencing an unbearably high amount of pain).
  Lower scores provide a better outcome for the patient as they are experiencing less pain post-operatively.
Time Frame: post-operative day 3
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 6 [4 to 8] | 4 [1 to 7]

2. Primary Outcome: Visual-analogue Pain Scale
Description: as for outcome 1
Time Frame: post-operative day 7
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 6 [3 to 9] | 4.1 [1 to 7]

3. Primary Outcome: Visual-analogue Pain Scale
Description: as for outcome 1
Time Frame: post-operative day 14
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 2.8 [1 to 5] | 3.56 [1 to 6]

4. Primary Outcome: Visual-analogue Anxiety Scale
Description: Visual-analogue anxiety scale is a tool used to measure anxiety intensity at a specific timepoint, asking a patient to use visuals to rate their current anxiety on a scale of 1 to 10.
  Results are reported as units on a scale, minimum 1 (experiencing the least amount of anxiety possible) to maximum of 10 (experiencing an unbearably high amount of anxiety).
  Lower scores provide a better outcome for the patient as they are experiencing less anxiety post-operatively.
Time Frame: post-operative day 3
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 4 [2 to 6] | 2.43 [1 to 6]

5. Primary Outcome: Visual-analogue Anxiety Scale
Description: as for outcome 4
Time Frame: post-operative day 7
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 4 [1 to 7] | 2.22 [1 to 5]

6. Primary Outcome: Visual-analogue Anxiety Scale
Description: as for outcome 4
Time Frame: post-operative day 14
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
Number analyzed (Participants) | 5 | 14
units on a scale | 2 [1 to 3] | 2.44 [1 to 6]

ADVERSE EVENTS:
Time Frame: 1 YEARS, 3 MONTHS
Arm/Group | Receiving Ropivacaine | Receiving Liposomal Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/14
Other Adverse Events (participants affected / at risk) | 0/5 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04801368/Prot_SAP_000.pdf